CLINICAL TRIAL: NCT07256158
Title: PET Guided Dose Reduction for InvOlved Site Radiotherapy In Early sTage Unfavourable Hodgkin Lymphoma: a Randomized, Phase III, Non-inferiority studY (PRIORITY Study)
Brief Title: PET Guided Dose Reduction for InvOlved Site Radiotherapy In Early sTage Unfavourable Hodgkin Lymphoma
Acronym: FIL_PRIORITY
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIL_PRIORITY
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin lymphoma; Early stage; unfavourable; untreated; ABVD; chemotherapy; radiotherapy; 20 Gy; 30 Gy; randomization; PET guided; involved site
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Intervention Model Description: Randomized, Phase III, Non-inferiority study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm - 20 Gy Radiotherapy (Experimental): Involved site radiotherapy (ISRT) Total dose of 20 Gy is administered in 10 daily fractions of 2.0 Gy, five times a week over 2 weeks
  Interventions: Radiation: 20 Gy Involved site radiotherapy
- Comparator arm - 30 Gy Radiotherapy (Active Comparator): Involved site radiotherapy (ISRT) Total dose of 30 Gy is administered in 15 daily fractions of 2.0 Gy, five times a week over 3 weeks
  Interventions: Radiation: 30 Gy Involved site radiotherapy

INTERVENTIONS:
Radiation: 20 Gy Involved site radiotherapy — Total dose 20 Gy Involved site radiotherapy
  Arms: Experimental arm - 20 Gy Radiotherapy
Radiation: 30 Gy Involved site radiotherapy — Total dose 30 Gy Involved site radiotherapy
  Arms: Comparator arm - 30 Gy Radiotherapy

SUMMARY:
The final analysis of GHSG HD11 study (not PET driven) showed that 30 Gy IFRT still remains the standard dose after 4 ABVD.

Early PET negativity might allow safe radiation de-escalation in patients achieving a metabolic complete response after 2 ABVD.

The aim of Priority trial is to explore whether radiotherapy could be safely deescalated to 20 Gy without loss of efficacy in patients treated with four cycles of ABVD who achieved complete metabolic response after the first two cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Histologically confirmed classical HL stage I, II unfavorable according to GHSG criteria;
* Patient with any nodal mass ≥ than 10 cm can be included
* No previous treatment for Hodgkin lymphoma;
* ECOG performance status 0 to 2;
* Presence of FDG-avid lymphoma lesions on baseline PET scan;
* Subject understands and voluntarily signs the informed consent form approved by the Independent Ethics Committee (IEC), prior to the initiation of any screening or study-specific procedures;
* Adequate organ and marrow function as defined below:

  * absolute neutrophil count > 1.0 x109/L
  * platelet count > 75 x109/L
  * Total bilirubin < 2 mg/dl without a pattern consistent with Gilbert's syndrome
  * Aspartate Transaminase and Alanine Transaminase (AST/ALT) < 3.0 X institutional Upper Limits of Normality (ULN)
  * Creatinine within normal institutional limits or creatinine clearance > 50 mL/min
* Women of childbearing potential must agree to use a highly effective method of contraception (oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device) from the signature of informed consent until six months after the last dose of treatment;
* Men must agree to use a highly effective method of contraception (barrier contraception or abstinence, when this is in line with the usual lifestyle of the subject) from the signature of informed consent until six months after the last dose of treatment;
* Women of childbearing potential must have a negative serum pregnancy test at screening.

Exclusion Criteria:

* Patients who meet any of the following criteria are not eligible to enroll:
* Stage II B- III- IV
* Hodgkin Lymphoma as "composite lymphoma" or nodular lymphocyte prevalence histological subtype
* Active HBV and HCV infection
* HIV seropositivity
* Pre-treatment with chemotherapy or radiation therapy
* Malignant disease within the last 5 years (excluding basal skin tumors and carcinoma in situ of the cervix)
* Women who are pregnant or breast feeding
* Absence of FDG-avid lymphoma lesions on baseline PET scan
* Significant history of neurologic, psychiatric, endocrinological, metabolic, immunologic, or hepatic disease that would preclude participation in the study or compromise ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2033-03-01 (Estimated); Study Completion 2033-03-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate if de-escalated ISRT dose (20 Gy) is not inferior to conventional ISRT dose (30 Gy) in terms of PFS in patients with newly diagnosed early-stage unfavourable HL achieving a complete metabolic response (DS 1-3) after 2 ABVD cycle | From the date of randomization to documented relapse, progression or to the patient's death as a result of any causes (up to 82 months).
  Progression-Free Survival (PFS) of the randomized population. Subjects with incomplete follow-up or with no disease evaluation will be censored at the date of last available documented status of freedom from failure.

SECONDARY OUTCOMES:
To compare OS rates between de-escalated ISRT dose (20 Gy) and conventional ISRT dose (30 Gy) in patients with newly diagnosed early-stage unfavourable HL achieving a complete metabolic response (DS 1-3) after 2 ABVD cycles; | From the time of randomization to death from any cause (up to 82 months)
  Overall Survival (OS) for the randomized population
To evaluate PFS for the whole population | From the date of consent to documented relapse, progression or death from any cause (up to 84 months)
  Progression free survival for the whole enrolled population
To evaluate OS for the whole population | From the date of consent to death from any cause (up to 84 months)
  Overall Survival (OS) for the whole population
To describe pattern of failure "in field", "marginal field", "out of field" relapse after conventional and reduced ISRT; | From the date of consent to death from any cause (up to 84 months)
  Incidence and severity of Adverse Events, graded according to the latest version of the Common Terminology Criteria for Adverse Events (CTCAE v 5.0) during the treatment
To report details on RT treatment volumes and dose distributions and to estimate the dose received by the organs at risk (OARs) in the two treatment arms | At time of radiotherapy (about 4 months from chemotherapy start)
  RT dose received by organs at risk (OARs).

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Ricardi, MD, Principal Investigator — SC Radioterapia U - AOU Città della Salute e della Scienza di Torino
Locations (38):
- Italy (38):
  - A.O.U. SS. Antonio e Biagio e C. Arrigo - S.C.D.U. Ematologia, Alessandria
  - A.O.R.N. G Moscati - U.O.C. Ematologia e Terapie cellulari avanzate, Avellino
  - IRCCS Centro Riferimento Oncologico - S.O.C. Oncologia medica e dei tumori immuno-correlati, Aviano
  - ASST Papa Giovanni XXIII - S.C. Ematologia, Bergamo
  - Clinica Humanitas Gavazzeni - U.O. Oncologia Medica, Bergamo
  - ASST Spedali Civili - S.C. Ematologia, Brescia
  - ARNAS "Brotzu" P.O. Businco - S.C. Ematologia e TMO, Cagliari
  - I.R.C.C.S. Istituto di Candiolo - FPO, Candiolo
  - ARNAS Garibaldi - U.O.C. Ematologia, Catania
  - A.O. S. Croce e Carle - S.C. Ematologia, Cuneo
  - A.S.L. Toscana Centro - SOC Oncoematologia, Florence
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - IRCCS Policlinico S. Martino - U.O. Ematologia e terapie cellulari, Genova
  - ASL Latina Ospedale S. Maria Goretti - UOC Ematologia con trapianto, Latina
  - ASST Grande Ospedale Metropolitano Niguarda - S.C. Ematologia, Milan
  - IRCCS Fondazione Istituto Nazionale Tumori - S.C. Ematologia, Milan
  - A.O.U. Ospedale Maggiore della Carità - S.C.D.U. Ematologia, Novara
  - A.O.U. di Padova - U.O.C. Ematologia, Padua
  - I.R.C.C.S. Istituto Oncologico Veneto - U.O.C. Oncologia 1, Padua
  - A.O. Ospedali Riuniti Villa Sofia-Cervello - Divisione di Ematologia, Palermo
  - IRCCS Fondazione Policlinico S. Matteo - S.C. Ematologia 1, Pavia
  - A.O. Ospedale S. Maria della Misericordia - Ematologia, Perugia
  - AUSL di Piacenza Ospedale Guglielmo da Saliceto - U.O.C. Ematologia e centro trapianti, Piacenza
  - AUSL di Ravenna Osp. S. Maria delle Croci - U.O.C. Ematologia, Ravenna
  - AUSL IRCCS Arcispedale S. Maria Nuova - S.C. Ematologia, Reggio Emilia
  - A.O.U. Policlinico Umberto I - U.O.C Ematologia, Roma
  - A.O.U. Sant'Andrea - U.O.C. Ematologia, Roma
  - Fondazione Policlinico Campus Bio-Medico - U.O.C. Ematologia e trapianto di cellule staminali, Roma
  - IRCCS Humanitas - U.O. Ematologia, Rozzano
  - IRCCS Fondazione Casa Sollievo della Sofferenza - UOC Ematologia e Trapianto di Cellule Staminali Ematopoietiche, San Giovanni Rotondo
  - A.O.U. Senese - U.O.C. Ematologia, Siena
  - A.O. Santa Maria - S.C. Oncoematologia, Terni
  - A.O.U. Città della Salute e della Scienza di Torino - S.C. Ematologia U, Torino
  - A.O.U. Città della Salute e della Scienza di Torino - S.C. Ematologia, Torino
  - ULSS 2 Ospedale Ca' Foncello - U.O.C. Ematologia, Treviso
  - A.S.U. Giuliano Isontina - S.C. Ematologia, Trieste
  - A.S.U. Friuli Centrale - Clinica Ematologica, Udine
  - A.O.U.I. di Verona - U.O.C. Ematologia, Verona

IPD SHARING:
Plan to Share IPD: Undecided